CLINICAL TRIAL: NCT06018129
Title: A Phase 1/2a, Open-Label, Dose Escalation Trial of GEN3017 With Expansion Cohorts in Relapsed or Refractory CD30+ Classical Hodgkin Lymphoma and CD30+ Non-Hodgkin Lymphoma
Brief Title: A First-in-human Trial of GEN3017 in Hodgkin Lymphoma and Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Genmab discontinued GEN3017 program following a strategic re-evaluation of Genmab's portfolio.
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT3017-01; 2023-503348-15-00 (EU CTIS Number); jRCT2031230576 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Classical Hodgkin Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- R/R CD30+ cHL Cohort (Experimental)
  Interventions: Biological: GEN3017
- R/R CD30+ TCL Cohort (Experimental)
  Interventions: Biological: GEN3017

INTERVENTIONS:
Biological: GEN3017 — Subcutaneous injection
  Other Names: DuoBody® CD3xCD30

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, immunogenicity, pharmacokinetics (PK), pharmacodynamics (PD), and anti-tumor activity of GEN3017 as a monotherapy in participants with relapsed or refractory (R/R) CD30-expressing lymphomas.

GEN3017 will be administered via subcutaneous injections.

All participants will receive active drug; no one will be given placebo.

DETAILED DESCRIPTION:
This multicenter trial will be conducted in 2 parts: Dose Escalation (phase 1) and Expansion (phase 2a).

The Dose Escalation Part (phase 1) of the trial will evaluate dose-limiting toxicities (DLTs) to determine the recommended phase 2 dose (RP2D), and if reached, the maximum tolerated dose (MTD) for R/R CD30+ classical Hodgkin lymphoma (cHL) and R/R CD30+ T-cell lymphoma (TCL), respectively.

The Expansion Part (phase 2a) will evaluate the anti-tumor activity of GEN3017 at the RP2D and selected dosage(s) will be assessed together with safety, immunogenicity, pharmacokinetics, and pharmacodynamics in R/R CD30+ cHL participants (including adults; and adolescent and young adults) and in participants with selected R/R CD30+ TCL subtypes (adults only).

ELIGIBILITY:
Key Inclusion Criteria:

Dose Escalation Part:

1. Must be at least 18 years of age. For participants in the R/R cHL Cohort in the United States (US) and Australia, must be at least 16 years of age.
2. Histologically confirmed R/R cHL or R/R TCL.
3. Participants must have at least 1 measurable lesion by fluorodeoxyglucose-positron emission tomography (FDG-PET) scan demonstrating positive lesion compatible with computed tomography (CT)- or magnetic resonance imaging (MRI)-defined anatomical tumor sites and a CT scan (or MRI) with involvement of ≥1 measurable nodal lesion and/or ≥1 measurable extranodal lesion.
4. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 for participants 18 years of age and above. For participants ≥16 and <18 years of age (US and Australia only), Karnofsky score of >60% per Karnofsky performance scale.
5. Confirmed CD30-positivity in tumor biopsy prior to the first dose of GEN3017.
6. R/R cHL Cohort:

   * Must have relapsed or progressive cHL after receiving at least 2 or 3 prior lines of therapy; OR
   * Refractory to the second line of therapy.

Key Exclusion Criteria:

1. Primary central nervous system (CNS) tumor or known CNS involvement.
2. Received prior investigational CD30-targeting therapy (except brentuximab vedotin).
3. Autologous hematopoietic stem cell transplant (HSCT) within 60 days (applies to both cHL and TCL). Allogeneic HSCT within 90 days (applies to cHL) prior to the first dose of GEN3017.
4. Chemotherapy within 2 weeks or major surgery within 4 weeks prior to the first dose of GEN3017.
5. Curative radiotherapy within 4 weeks or palliative radiotherapy within 2 weeks prior to the first dose of GEN3017.
6. Treatment with an investigational drug within 4 weeks or 5 half-lives of the drug, whichever is shorter prior to the first dose of GEN3017 or currently receiving any other investigational agents.
7. Prior treatment with live, attenuated vaccines within 30 days prior to the first dose of GEN3017.
8. Receiving immunosuppressive drugs or systemic corticosteroids such as prednisone at doses >25 milligrams (mg) daily or its equivalent within 14 days prior to the first dose of GEN3017.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (4):
- United States (3):
  - City of Hope Helford Clinical Research Hospital, Duarte, California
  - Washington University School of Medicine, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas
- Peter MacCallum Cancer Institute trading as Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results Summary in Plain Language — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-503348-15-00

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was conducted in participants with classical Hodgkin lymphoma and T-cell lymphoma. This trial was planned to be conducted in 2 parts: dose escalation and expansion; however, it was terminated during dose escalation and did not proceed to expansion.
Groups:
- GEN3017 Medium Priming Dose + Low Full Dose: Participants received GEN3017 at a medium priming dose and a low full dose.
- GEN3017 High Priming Dose + High Full Dose: Participants received GEN3017 at a high priming dose and a high full dose.
- GEN3017 Low Priming Dose + High Full Dose: Participants received GEN3017 at a low priming dose and a high full dose.
Period: Overall Study
Arm/Group | GEN3017 Medium Priming Dose + Low Full Dose | GEN3017 High Priming Dose + High Full Dose | GEN3017 Low Priming Dose + High Full Dose
Started | 3 | 3 | 3
Received At Least 1 Dose of Trial Treatment | 3 | 3 | 3
Number of Participants Enrolled With Classical Hodgkin Lymphoma | 1 | 3 | 0
Number of Participants Enrolled With T-cell Lymphoma | 2 | 0 | 3
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 3
Not completed — Death | 1 | 1 | 2
Not completed — Sponsor Decision | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Measured in the Full Analysis Set (FAS), which included participants enrolled and treated with at least 1 dose of GEN3017.
Groups:
- Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose; T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose: Participants received GEN3017 at a medium priming dose and a low full dose.
- Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose: Participants received GEN3017 at a high priming dose and a high full dose.
- T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose: Participants received GEN3017 at a low priming dose and a high full dose.
- Total: Total of all reporting groups
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose | Total
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 | 62.0 (17.3) | 40.0 (19.8) | 56.0 (27.9) | 52.8 (20.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 1 | 1 | 1 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Missing | 0 | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 1 | 2 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian Indian | 0 | 0 | 0 | 0 | 0
  Asian Other | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  Chinese | 0 | 0 | 0 | 0 | 0
  Japanese | 0 | 0 | 0 | 0 | 0
  Malay | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following toxicities except those that were clearly due to the underlying disease or extraneous cause: all Grade 5 toxicities, hematological toxicities (Grade 4 neutropenia, Grade 3 and Grade 4 febrile neutropenia lasting >2 days, Grade 4 thrombocytopenia of any duration with clinically significant bleeding or ≥ Grade 3 thrombocytopenia requiring platelet transfusion, Grade 4 anemia), non-hematological toxicities (Grade 4 cytokine release syndrome [CRS] per American Society for Transplantation and Cellular Therapy [ASTCT] criteria or Grade 3 unresolved to ≤ Grade 2 within 48 hours following adequate intervention, Grade 4 immune effector cell-associated neurotoxicity syndrome [ICANS] according to ASTCT criteria or Grade 3 unresolved to ≤ Grade 2 within 48 hours following adequate intervention, tumor lysis syndrome [TLS] Grade 4 or Grade 3 unresolved within 5 days, any ≥ Grade 3 [severe or life-threatening] non-hematological toxicities [with exceptions]).
Time Frame: 21 days
Population: Measured in the Dose-Determining Set, which included all participants from the Safety Set who met the minimum exposure criteria and had either completed the DLT observation period or had experienced a DLT during the specified time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 1 | 3
Participants | 0 | 2 | 0 | 0

2. Primary Outcome: Dose Escalation Part: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE was therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: Up to approximately 1 year 2 months
Population: Measured in the Safety Set, which included participants enrolled and treated with at least 1 dose of GEN3017.
Measure: Count of Participants; unit: Participants
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
Participants | 1 | 3 | 2 | 3

3. Secondary Outcome: Dose Escalation Part: Maximum (Peak) Plasma Concentration (Cmax) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: Measured in the Pharmacokinetic (PK) Analysis Set, which included all participants who received at least 1 dose of GEN3017 and provided at least 1 evaluable PK sample. As pre-specified, data were collected and are reported per Classical Hodgkin Lymphoma and T cell Lymphoma groups. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected and data were collected and are reported for the dose escalation part only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
micrograms per milliliter (ug/mL)
  Day 1 | 0.0064 | 0.0449 (30.4032) | 0.0025 (148.0402) | 0.0005 (NA) — Geometric coefficient of variation (Geo CV%) could not be calculated because all reported values were identical, resulting in a geometric standard deviation of 1. As a consequence, the Geo CV% could not be calculated.
  Day 8 | 0.0389 | 0.2503 (15.7057) | 0.0056 (142.6003) | 0.0063 (33.1330)

4. Secondary Outcome: Dose Escalation Part: Time to Reach Cmax (Tmax) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: Measured in the PK Analysis Set, which included all participants who received at least 1 dose of GEN3017 and provided at least 1 evaluable PK sample. As pre-specified, data were collected and are reported per Classical Hodgkin Lymphoma and T cell Lymphoma groups. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected and data were collected and are reported for the dose escalation part only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
days
  Day 1 | 2.6069 | 6.6736 (164.5774) | 1.6424 (95.0650) | 0.2322 (0.9590)
  Day 8 | 3.0340 | 3.8858 (51.7969) | 2.2907 (18.1691) | 2.0079 (75.6204)

5. Secondary Outcome: Dose Escalation Part: Pre-dose (Trough) Concentration (Ctrough) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: While blood samples were collected to derive data for this planned PK outcome measure, the study was terminated prior to that data being generated, analyzed, summarized, or made available by the study sponsor. Therefore, no PK data can be presented here. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected.
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Dose Escalation Part: Area Under the Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: as for outcome 5
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Dose Escalation Part: Area Under the Concentration-time Curve (AUC) From Time Zero to Last Quantifiable Sample (AUClast) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
day*ug/mL
  Day 1 | 0.0375 | 0.3642 (56.7248) | 0.0122 (132.1774) | 0.0034 (2.2752)
  Day 8 | 0.1798 | 1.2989 (22.6968) | 0.0282 (160.8826) | 0.0304 (30.4785)

8. Secondary Outcome: Dose Escalation Part: Elimination Half-life (T1/2) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: as for outcome 5
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Dose Escalation Part: Total Body Clearance (CL) of Drug From Plasma of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: as for outcome 5
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Dose Escalation Part: Volume of Distribution (Vd) of GEN3017
Description: Venous blood samples were collected for analyzing concentrations of GEN3017.
Time Frame: Day 1 and Day 8
Population: as for outcome 5
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Dose Escalation Part: Number of Participants With Anti-drug Antibodies (ADAs) to GEN3017
Description: Venous blood samples were drawn for analysis of ADAs in serum samples.
Time Frame: Up to approximately 1 year 2 months
Population: Measured in the Immunogenicity Analysis Set, which included all participants who received at least 1 dose of GEN3017 and had a baseline and at least 1 evaluable on-treatment ADA sample. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected and data were collected and are reported for the dose escalation part only.
Measure: Count of Participants; unit: Participants
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
Participants | 0 | 1 | 1 | 0

12. Secondary Outcome: Dose Escalation Part: Objective Response Rate (ORR)
Description: ORR was defined as the number of participants with a best overall response of complete response (CR) or partial response (PR) based on the Lugano criteria as assessed by investigator. All other categories, including not evaluable, were considered non-response. CR was defined as all of the following: disappearance of all target and non-target tumor lesions, and reduction in short axis to <10 millimeters (mm) in all pathological target and non-target lymph nodes, and normalization of tumor marker level (if applicable). PR was defined as ≥30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Data are presented for the number of participants with ORR.
Time Frame: Up to approximately 1 year 2 months
Population: Measured in the FAS, which included participants enrolled and treated with at least 1 dose of GEN3017. As pre-specified, data were collected and are reported per Classical Hodgkin Lymphoma and T cell Lymphoma groups. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected and data were collected and are reported for the dose escalation part only.
Measure: Count of Participants; unit: Participants
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 1 | 3 | 2 | 3
Participants | 0 | 1 | 1 | 0

13. Secondary Outcome: Dose Escalation Part: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of response (CR or PR) to the date of progressive disease or death, whichever occurred earlier based on the Lugano criteria as assessed by investigator.
Time Frame: Up to approximately 1 year 2 months
Population: Measured in the FAS, which included participants enrolled and treated with at least 1 dose of GEN3017, in participants who achieved a response. As pre-specified, data were collected and are reported per Classical Hodgkin Lymphoma and T cell Lymphoma groups. The trial was terminated prior to the start of the expansion part. Therefore, no data for the expansion part were collected and data were collected and are reported for the dose escalation part only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 1 | 1 | 0
months |  | 2.23 [NA to NA] — Data could not be calculated as there was only 1 participant with a response. | 4.17 [NA to NA] — Data could not be calculated as there was only 1 participant with a response. |

14. Secondary Outcome: Dose Escalation Part: Time to Response (TTR)
Description: TTR was defined as the time from Day 1 to first documentation of objective response (CR or PR) in participants achieving PR or CR based on the Lugano criteria as assessed by investigator.
Time Frame: Up to approximately 1 year 2 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
Number analyzed (Participants) | 0 | 1 | 1 | 0
months |  | 1.18 (NA) — Data could not be calculated as there was only 1 participant with a response. | 1.25 (NA) — Data could not be calculated as there was only 1 participant with a response. |

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year 2 months
Description: Measured in the Safety Analysis Set, which included participants enrolled and treated with at least 1 dose of GEN3017.
Arm/Group | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/3 | 1/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 2/2 | 2/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose (N=1) | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose (N=3) | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose (N=2) | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose (N=3)
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Classical Hodgkin Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose (N=1) | Classical Hodgkin Lymphoma: GEN3017 High Priming Dose + High Full Dose (N=3) | T-cell Lymphoma: GEN3017 Medium Priming Dose + Low Full Dose (N=2) | T-cell Lymphoma: GEN3017 Low Priming Dose + High Full Dose (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Strongyloides test positive (Investigations) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Injection site reaction (General disorders) | 1 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination meant only a small number of participants were analyzed and data were not collected for the dose expansion part.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT06018129/Prot_SAP_000.pdf